CLINICAL TRIAL: NCT02903381
Title: Phase II Trial of the PD-1 Antibody Nivolumab in Combination With Lenalidomide and Low Dose Dexamethasone in Patients With High-Risk Smoldering Multiple Myeloma
Brief Title: A Phase II Trial If Nivolumab, Lenalidomide and Dexamethasone in High Risk Smoldering Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Bristol-Myers Squibb (Industry); Multiple Myeloma Research Consortium (Network); Blood Cancer Research Partnership (Other)
Responsible Party: Principal Investigator, Irene Ghobrial, MD, Prinicipal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-242; CA209-607 (Other: Bristol-Myers Squibb)
Record Dates: First submitted 2016-08-30; First posted 2016-09-16 (Estimated); Results first posted 2023-06-13 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-05

CONDITIONS: Smoldering Multiple Myeloma
Keywords: Smoldering Multiple Myeloma
MeSH Terms: conditions — Smoldering Multiple Myeloma | interventions — Nivolumab; Lenalidomide; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nivolumab, Lenalidomide, Dexamethasone (Experimental): * A treatment cycle is defined as 28 consecutive days.
  * Participants will receive 6 cycles of induction therapy followed by 6 cycles of maintenance therapy with lower doses of lenalidomide and no dexamethasone for a total of 12 months.
  Interventions: Drug: Nivolumab; Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Nivolumab — Intravenous, predetermined dosage, Days 1 and 15 during cycles 1-12 and
  Other Names: Opdivo®
Drug: Lenalidomide — Oral, predetermined dosage, Days 1-21 of cycle 1-12
  Other Names: Revlimid
Drug: Dexamethasone — Oral, Days 1, 8, 15 of cycle 1-6
  Other Names: Decadron; Dexasone; Diodex; Hexadrol; Maxidex

SUMMARY:
This research study is evaluating a new drug called "nivolumab" as a possible treatment for smoldering multiple myeloma in order to prevent or postpone development of active multiple myeloma.

- Patients with smoldering multiple myeloma do not have symptoms but are at risk for progressing to active multiple myeloma. Multiple myeloma is a cancer of the plasma cell, which is an important part of the immune system. Patients with active multiple myeloma generally require treatment.

DETAILED DESCRIPTION:
* This research study is a Phase II clinical trial, which tests the effectiveness of an investigational drug(s). The investigational drugs used in this research study are;

  * nivolumab
  * lenalidomide
  * dexamethasone.
* Preliminary experience suggests that the combination of lenalidomide and dexamethasone may prevent or postpone smoldering multiple myeloma (SMM) from becoming active multiple myeloma. The purpose of this research study is to determine if the addition of nivolumab may improve the rate of prevention in combination with lenalidomide and dexamethasone.
* "Investigational" means that the FDA (the U.S. Food and Drug Administration) has not approved the combination of nivolumab, lenalidomide and dexamethasone as a treatment regimen.
* Lenalidomide is an immunomodulatory drug derived from thalidomide. Lenalidomide works by stopping blood flow to your cancer cells and signaling your cancer cells to die off. The FDA has approved lenalidomide for the treatment of many types of cancer including multiple myeloma, and myelodysplastic syndromes.
* Dexamethasone, also FDA approved, is a type of steroid and is usually combined with other chemotherapy for the treatment of blood cancers, such as myeloma and leukemias.
* Nivolumab is approved by the FDA for some lung cancers, some skin cancers, some kidney cancers, and Hodgkin lymphoma. It is currently being evaluated for use in the treatment of several other types of cancers. Nivolumab may kill or stop cancer cells from growing by blocking a signal in the cells allowing the immune system to fight the cancer. This drug is a human monoclonal antibody, which is a molecule that is made in a laboratory that is designed to act identically to cells in the immune system.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years.
* Must meet criteria of high risk smoldering MM based on the criteria described below:

  -- Definition of high-risk SMM:

  --- Bone marrow clonal plasma cells ≥10% and ≤60% and any one or more of the following:
  * Serum M protein ≥3.0g/dL (IgA, IgG, IgM, or IgD)
  * IgA SMM
  * Immunoparesis with reduction of two uninvolved immunoglobulin isotypes
  * Serum involved/uninvolved free light chain ratio ≥8 (but less than 100)

    ----- Free Light Chain Smoldering Myeloma patients as defined in section 2.4 are not excluded
  * Progressive increase in M protein level (Evolving type of SMM)

    ----- Increase in serum monoclonal protein by ≥10% on two successive evaluations within a 6 month period
  * Bone marrow clonal plasma cells 50-60%
  * Abnormal plasma cell immunophenotype (≥95% of bone marrow plasma cells are clonal) and reduction of one or more uninvolved immunoglobulin isotypes
  * t (4;14) or del 17p or 1q gain
  * Increased circulating plasma cells
  * MRI with diffuse abnormalities or 1 focal lesion
  * PET-CT with one focal lesion with increased uptake without underlying osteolytic bone destruction
  * Urine monoclonal light chain excretion ≥500 mg/24 hours
* ECOG Performance Status (PS) 0, 1, or 2 (Appendix A)
* The following laboratory values obtained 21 days prior to registration and confirmed prior to the first dose of study drug:

  * ANC ≥1000/ µL
  * PLT ≥ 50,000/µL. Platelet transfusions to help patients meet eligibility criteria are not allowed within 3 days before study enrollment.
  * Total bilirubin ≤ 1.5 mg/dL (If total is elevated check direct and if normal patient is eligible.)
  * AST ≤ 3 x institutional upper limit of normal (ULN)
  * ALT ≤ 3 x institutional upper limit of normal (ULN)
  * Creatinine ≤ 1.5 mg/dL
  * WBC ≥2000/μL
* Ability to understand and willingness to sign a written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
* Female patients who are postmenopausal for at least 1 year before the screening visit or are surgically sterile. Females of childbearing potential* must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 10 - 14 days and again within 24 hours prior to prescribing lenalidomide for Cycle 1 (prescriptions must be filled within 7 days as required by Revlimid REMS®) and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide. Females of reproductive potential must agree to follow instructions for method(s) of contraception for the duration of treatment with any study drug(s) plus 5 half-lives of study plus 30 days (duration of ovulatory cycle) for a total of 120 days post treatment completion. Women must not breastfeed. -- A female of childbearing potential is a sexually mature female who:

  * Has not undergone a hysterectomy (the surgical removal of the uterus) or bilateral oophorectomy (the surgical removal of both ovaries) or
  * Has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time during the preceding 24 consecutive months)
* All study participants must be registered into the mandatory Revlimid REMS® program, and be willing and able to comply with the requirements of the REMS® program.
* Females of reproductive potential must adhere to the scheduled pregnancy testing as required in the Revlimid REMS® program.
* Men must agree to use a latex condom during sexual contact with a female of childbearing potential even if they have had a successful vasectomy during the entire study treatment period and through 154 days after the last dose of study drug or agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [eg, calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception.)

Exclusion Criteria:

* No evidence of CRAB criteria* or new criteria of active MM which including the following:

  * Increased calcium levels (corrected serum calcium >0.25 mmol/dL above the upper limit of normal or >.275 mmol/dL) related to MM
  * Renal insufficiency (attributable to MM)
  * Anemia (Hb 2g/dL below the lower limit of normal or <10g/dL) related to MM
  * Bone lesions (lytic lesions or generalized osteoporosis with compression fractures)
  * Bone marrow plasma cells ≥60%
  * Serum involved/uninvolved FLC ratio ≥100, provided the absolute level of the involved free light chain is at least 100 mg/L and repeated twice (light chain smoldering myeloma as described in section 2.4 is not an exclusion criteria).
  * MRI with two or more focal lesions that are at least 5 mm or greater in size --- *Participants with CRAB criteria that are attributable to conditions other than the disease under study may be eligible
* Other concurrent chemotherapy, immunotherapy, radiotherapy, or any ancillary therapy considered investigational. Prior therapy with bisphosphonate is allowed. Prior therapy for smoldering myeloma MM may not be an exclusion criterion, discussion with Principal Investigator must occur before enrolling patients with prior treatments. Prior radiation therapy to a solitary plasmacytoma is allowed.
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
* Diagnosed or treated for another malignancy within 2 years of enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low-risk prostate cancer after curative therapy.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Autoimmune disease: Patients with a history of inflammatory bowel disease, including ulcerative colitis and Crohn's Disease, are excluded from this study, as are patients with a history of symptomatic disease (eg, rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, autoimmune pneumonitis, autoimmune vasculitis [eg, Wegener's Granulomatosis]) and motor neuropathy considered of autoimmune origin (e.g. Guillain-Barre Syndrome and Myasthenia, Gravis). Patients with Hashimoto's thyroiditis are eligible to go on study.
* Pregnant or nursing women will be excluded from the study because lenalidomide is an agent with the potential for teratogenic or abortifacient effects.
* History of severe allergic reactions attributed to compounds of similar chemical or biologic composition to Nivolumab or lenalidomide.
* Known seropositive for or active viral infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV). Patients who are seropositive because of hepatitis B virus vaccine are eligible.
* Major surgery within 4 weeks before enrollment.
* Myeloma-related central nervous system involvement.
* Known Amyloid involvement.
* Participation in other clinical trials, including those with other investigational agents not included in this trial, within 30 days of the start of this trial and throughout the duration of this trial.
* Prior CVA with persistent neurological deficit.
* Inability to tolerate thromboprophylaxis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-10-20 (Actual); Primary Completion 2018-06-28 (Actual); Study Completion 2021-09-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Irene M. Ghobrial, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Nivolumab, Lenalidomide, Dexamethasone: * A treatment cycle is defined as 28 consecutive days.
  * Participants will receive 6 cycles of induction therapy followed by 6 cycles of maintenance therapy with lower doses of lenalidomide and no dexamethasone for a total of 12 months.
  Nivolumab: Intravenous, predetermined dosage, Days 1 and 15 during cycles 1-12 and
  Lenalidomide: Oral, predetermined dosage, Days 1-21 of cycle 1-12
  Dexamethasone: Oral, Days 1, 8, 15 of cycle 1-6
Period: Overall Study
Arm/Group | Nivolumab, Lenalidomide, Dexamethasone
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Ten patients were screened and completed baseline visits; however, two patients did not start protocol therapy and are excluded from demographic, safety, and clinical outcomes
Arm/Group | Nivolumab, Lenalidomide, Dexamethasone
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 3
Age, Continuous [Median (Full Range); unit: years] | 60 [49 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8
ECOG Performance Status [Count of Participants; unit: Participants]
  00 - Fully Active | 5
  01 - Restricted | 3

OUTCOME MEASURES:

1. Primary Outcome: 2 Year Progression Free Percent
Description: The primary endpoint will be the 2-year progression-free percent and will be reported with corresponding 90% confidence interval. All patients who have received one dose of study treatment will be included for the analysis, including those who die or are lost to follow-up before 2 years. Progression is defined as ≥ 25% increase and an absolute increase of ≥ 0.5g/dL from their nadir in their serum or urine m-spike or FLC with no CRAB features attributable to MM progression.
Time Frame: 2 Year
Population: All patients receiving any amount of protocol treatment. Patients who have progressed or lost to follow-up prior to two years are counted as failures; only patients followed and progression-free for at least two years are counted as successes.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Nivolumab, Lenalidomide, Dexamethasone
Number analyzed (Participants) | 8
percentage of participants | 62.5 [28.9 to 88.9]

2. Secondary Outcome: Objective Response Percent
Description: The percent of patients with objective response defined as achieving a partial response or better according to the modified International Myeloma Working Group (IMWG) criteria
Time Frame: 2 Years
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Nivolumab, Lenalidomide, Dexamethasone
Number analyzed (Participants) | 8
percentage of participants | 87.5 [52.9 to 99.4]

3. Secondary Outcome: Time to Progression Probability at 2-years
Description: Time to progression (TTP) is defined as the time from protocol therapy initiation until documented progression, censored at date last known progression-free for those who have not progressed, up to 24 months post initiation of therapy.
Time Frame: Baseline to documented progression, up to 24 months post initiation of therapy.
Measure: Number (90% Confidence Interval); unit: probability
Arm/Group | Nivolumab, Lenalidomide, Dexamethasone
Number analyzed (Participants) | 8
probability | 0.75 [0.54 to 1.0]

4. Secondary Outcome: Duration of Response Probability at 2-years
Description: Kaplan-Meier method, duration of response probability in patients with partial response or better. Events defined as confirmed progression or death from any cause
Time Frame: time from objective response to disease progression or death, or date last known progression-free and alive for those who have not progressed or died, up to 24 months post initiation of therapy.
Population: 7 of 8 patients achieved a confirmed objective response and are included in duration of response analysis
Measure: Number (90% Confidence Interval); unit: probability
Arm/Group | Nivolumab, Lenalidomide, Dexamethasone
Number analyzed (Participants) | 7
probability | 0.71 [0.48 to 1.0]

5. Secondary Outcome: Progression Free Survival (PFS) Probability at 2-years
Description: Kaplan-Meier method, percent of patients alive and progression-free at 2-years
Time Frame: Baseline to disease progression or death from any cause, censored at date last known progression free for those who have not progressed or died, up to 24 months post initiation of therapy.
Measure: Number (90% Confidence Interval); unit: probability
Arm/Group | Nivolumab, Lenalidomide, Dexamethasone
Number analyzed (Participants) | 8
probability | 0.75 [0.54 to 1.0]

6. Secondary Outcome: Overall Survival Probability at 2-years
Description: Kaplan-Meier method, percent alive at 2-years
Time Frame: Baseline to death or date last known alive, up to 24 months post initiation of therapy.
Measure: Number (90% Confidence Interval); unit: probability
Arm/Group | Nivolumab, Lenalidomide, Dexamethasone
Number analyzed (Participants) | 8
probability | 1.0 [1.0 to 1.0]

7. Secondary Outcome: Progression Free Survival Rate-Without Cyclophosphamide
Description: It is expected that approximately 20% of the patients will receive cyclophosphamide (CTX) for mobilization and this may influence the PFS. Therefore, in a secondary analysis the 2 year PFS rate will be evaluated among those patients who did not receive CTX.
Time Frame: 2 Years
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Nivolumab, Lenalidomide, Dexamethasone
Number analyzed (Participants) | 7
percentage of participants | 71.4 [48.2 to 100]

8. Secondary Outcome: Number of Participants With Adverse Events
Description: For toxicity reporting, all adverse events and laboratory abnormalities will be graded and analyzed using CTCAE version 4 as appropriate.
Time Frame: Baseline to 2 Years
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab, Lenalidomide, Dexamethasone
Number analyzed (Participants) | 8
Participants | 8

ADVERSE EVENTS:
Time Frame: Adverse Events or toxicity events assessed/monitored from the day of consent up to end of treatment visit for an average of 14 months. All-Cause Mortality as well as Serious Adverse Events were assessed up to 4.5 years.
Description: Toxicity assessments performed on day 1 of cycles 1-12 (each cycle is 28 days); additional assessment on end-of-treatment visit. Reported toxicities have either "definite," "probable," or "possible" attribution to any of protocol treatments.
Arm/Group | Nivolumab, Lenalidomide, Dexamethasone
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 1/8
Other Adverse Events (participants affected / at risk) | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nivolumab, Lenalidomide, Dexamethasone (N=8)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nivolumab, Lenalidomide, Dexamethasone (N=8)
Fatigue (General disorders) | 6 (9)
Neutrophil count decreased (Investigations) | 6 (21)
Anemia (Blood and lymphatic system disorders) | 5 (14)
Hypophosphatemia (Metabolism and nutrition disorders) | 5 (10)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 (7)
White blood cell decreased (Investigations) | 5 (14)
Constipation (Gastrointestinal disorders) | 4 (7)
Edema limbs (General disorders) | 4 (5)
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 (7)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (5)
Platelet count decreased (Investigations) | 4 (11)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Dizziness (Nervous system disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Hyperthyroidism (Endocrine disorders) | 3 (5)
Insomnia (Psychiatric disorders) | 3 (3)
Alanine aminotransferase increased (Investigations) | 2 (4)
Aspartate aminotransferase increased (Investigations) | 2 (4)
Blurred vision (Eye disorders) | 2 (2)
Creatinine increased (Investigations) | 2 (4)
Dysgeusia (Nervous system disorders) | 2 (2)
Flushing (Vascular disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (5)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2)
Hypothyroidism (Endocrine disorders) | 2 (2)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 2 (2) — Polydipsea, Psuedo Gout
Thromboembolic event (Vascular disorders) | 2 (2)
Blood bilirubin increased (Investigations) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Edema face (General disorders) | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 1 (1) — Visual Disturbances
Headache (Nervous system disorders) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1)
Laryngitis (Infections and infestations) | 1 (1)
Libido decreased (Psychiatric disorders) | 1 (1)
Localized edema (General disorders) | 1 (1)
Mucosal infection (Infections and infestations) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1) — Hyperactivity
Pain (General disorders) | 1 (1)
Periorbital edema (Skin and subcutaneous tissue disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Scalp pain (Skin and subcutaneous tissue disorders) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Superficial thrombophlebitis (Vascular disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-01-23): https://cdn.clinicaltrials.gov/large-docs/81/NCT02903381/Prot_SAP_000.pdf
  • Informed Consent Form (2019-05-07): https://cdn.clinicaltrials.gov/large-docs/81/NCT02903381/ICF_001.pdf